CLINICAL TRIAL: NCT01427348
Title: Maintaining the Head Extension by an Assistant Decreases Dental Contact Between Laryngoscope Blade and Maxillary Incisors During Direct Laryngoscopy
Brief Title: Maintaining the Head Extension by an Assistant Decreases Dental Contact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_dental injury
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Dental Contact During Direct Laryngoscopy
MeSH Terms: interventions — Dental Assistants

ARMS (2):
- with assistant (Experimental): head extension by an assistant during direct laryngoscopy
  Interventions: Procedure: with assistant
- without assistant (Active Comparator): without the help of an assistant during direct laryngoscopy
  Interventions: Procedure: without assistant

INTERVENTIONS:
Procedure: with assistant — head extension by an assistant during direct laryngoscopy
  Arms: with assistant
Procedure: without assistant — without head extension by an assistant during direct laryngoscopy
  Arms: without assistant

SUMMARY:
The purpose of this study is to determine whether the head extension by an assistant decreases dental contact between laryngoscope blade and maxillary incisors during direct laryngoscopy

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery that requires general anesthesia

Exclusion Criteria:

* disease or injury of cervical spine
* dentoalveolar injury
* history of difficult intubation
* anatomical anomaly of face or airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
dental contact | up to 10 minutes
  dental contact between laryngoscope blade and maxillary incisors

SECONDARY OUTCOMES:
teeth distance | up to 10 minutes
  teeth distance between laryngoscope blade and maxillary incisors

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Lee JM, Bahk JH. Assisted head extension minimizes the frequency of dental contact with laryngoscopic blade during tracheal intubation. Am J Emerg Med. 2013 Dec;31(12):1629-33. doi: 10.1016/j.ajem.2013.08.019. Epub 2013 Sep 14. PMID 24041638